CLINICAL TRIAL: NCT04774081
Title: Development of a Novel Method to Measure Insulin Sensitivity in Humans: A Pilot Study
Acronym: CGM-PEPTIDE
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Eric Ravussin, Boyd Professor, Associate Executive Director for Clinical Science, Pennington Biomedical Research Center
Other Study IDs: PBRC2020-009
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study group: Participants will be recruited among those whose insulin sensitivity has been previously measured by a high-dose euglycemic-hyperinsulinemic clamp at Pennington Biomedical during the last 5 years and indicated their wiliness to be re-contacted for future research
  Interventions: Device: 24h Continuous glucose monitoring and urinary C-peptide collection

INTERVENTIONS:
Device: 24h Continuous glucose monitoring and urinary C-peptide collection — Participants will be admitted to the research clinic for a 24-hour stay in a metabolic chamber. During the chamber stay, all urine excreted will be collected to assess C-peptide urinary excretion rate and interstitial glucose will be measured by a continuous glucose monitor (CGM). Participants will consume a eucaloric diet (50% carbohydrates, 30% fat and 20% protein).

SUMMARY:
This study will determine whether the ratio between 24h C-peptide urinary excretion rate and average 24h circulating glucose represent a good correlate of what is measured by the gold standard, i.e. M (glucose disposal rate) from a euglycemic-hyperinsulinemic clamp

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Age 18-65 y
* BMI between 20 kg/m2 and 35 kg/m2 (inclusive)
* Are willing to consume pre-prepared meals
* Have completed a high-dose (≥80 mIU/m2/min) euglycemic-hyperinsulinemic clamp during the last five years at Pennington Biomedical. The data from the previous PBRC clamp will be pulled and used in conjunction with data from this study.
* Willing to have blood and urine stored for future use

Exclusion Criteria:

* Major lifestyle changes since the euglycemic-hyperinsulinemic clamp was performed (i.e. gain/lost weight, stopped smoking, began/stop exercise).
* Unstable weight in the last 3 months [gain or loss >10 lb (or 4.5 kg)]
* Diagnosed with diabetes
* Untreated hypertension and average screening blood pressure >140/90 mmHg
* Previous bariatric surgery (or other surgeries) for obesity or weight loss
* Chronic use of medications affecting metabolism or sleep*
* History of neurological disease
* History of cardiovascular disease, or other chronic diseases, that might affect pancreatic or glucose metabolism.
* Pregnant, planning to become pregnant, or breastfeeding
* Adherence to special restrained diets (e.g., low-CHO, low-fat, or vegetarian/vegan diets) over the last 3 months. *Sporadic use of these medications is fine (however, enrollment will depend on a case-by-case basis). If taking sporadically, participants should not be taking the medication for 1-month prior to the first visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited among those whose insulin sensitivity has been previously measured by a high-dose euglycemic-hyperinsulinemic clamp at Pennington Biomedical during the last 5 years and indicated their wiliness to be re-contacted for future research
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Glycemia (Continuous Glucose Monitoring) | 24 hours
Urinary C-peptide | 24 hours

OTHER OUTCOMES:
M-value at a high-dose (≥80 mIU/m2/min) euglycemic-hyperinsulinemic clamp. | Up to 5 years before the CGM and C-peptide assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States